CLINICAL TRIAL: NCT03303443
Title: Empirical Mode Decomposition in the Electroencephalogram During General Anesthesia Between Generations
Brief Title: Empirical Mode Decomposition in the Electroencephalogram
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201508007RIN
Record Dates: First submitted 2015-12-01; First posted 2017-10-06 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2019-04

CONDITIONS: Depth of Anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Younger: 20-40 years old patients
- Elderly: over 60 years old patients

SUMMARY:
Bispectral index (BIS), a standard monitor for perioperative monitor of patient's conscious level, is a noninvasive medical technique for monitoring and recording the electrical activity of brain.

DETAILED DESCRIPTION:
The electroencephalogram and BIS data have lots of information. Fourier transformation to decompose EEG was first applied on the EEG signaling until now. The disadvantages of Fourier transformation is hard to deal with physical signals, which was modulated by autonomic system and factors. The Hilbert-Huang transform (HHT) was proposed to decompose EEG signal into intrinsic mode functions (IMF) since 2004. HHT can obtain instantaneous frequency data and work well for data that is nonstationary and nonlinear. HHT have been applied for wild ranges, not only in the analysis of arrhythmia for medical and public health fields, but also in the earthquake detection and earth physics detection…etc.

The relationship between frontal EEG patterns and general anesthesia remain poorly understood. It can only say that the increase in frontal EEG power and shift power to lower frequencies during general anesthesia from publications. The investigators are going to compare the EEG signal between generations, try to find the difference in aging using empirical mode decomposition method.

ELIGIBILITY:
Inclusion Criteria:

1. 20-40y/o or over 60y/o
2. Scheduled for low risk general anesthesia
3. Suitable for surgery after interviewed by anesthesiologist

Exclusion Criteria:

1. Not suitable for general anesthesia
2. High risk patient
3. Allergic to the EEG sensor

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20-40y/o patients or over 60y/o patients without severe systemic disease who were scheduled for general anesthesia.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
EEG power calculation | During the operation time.
  The investigator use root mean square energy to calculate EEG power.

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Fang Tsai, MD, Study Chair — National Taiwan University Hospital
Locations (1):
- Feng-Fang Tsai, Taipei, Taiwan